CLINICAL TRIAL: NCT01914913
Title: An Open Labeled Clinical Study to Evaluate the Safety and Efficacy OF Autologous Bone Marrow Derived Mono Nuclear Stem Cell (BMMNCs) in Retinitis Pigmentosa. It is Self Funded (Patients' Own Funding) Clinical Trial
Brief Title: Clinical Study to Evaluate Safety and Efficacy of BMMNC in Retinitis Pigmentosa
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chaitanya Hospital, Pune (Other)
Responsible Party: Principal Investigator, Dr. Sachin Jamadar, Co -investigator, Chaitanya Hospital, Pune
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSCC/BMRP/2013//01
Record Dates: First submitted 2013-07-31; First posted 2013-08-02 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Retinitis Pigmentosa
Keywords: retinitis pigmentosa; Bone marrow; stem cell; BMMNC
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BMMNCs (Other): BMMNCs
  Interventions: Biological: BMMNCs

INTERVENTIONS:
Biological: BMMNCs — Intervention therapy , Total 3 doses ,in 30 days ,in 7days interval ,transfer of Autologous Bone Marrow derived Mono Nuclear Stem Cell (BMMNCs)

SUMMARY:
Retinitis pigmentosa is an eye disease in which there is damage to the retina. The retina is the layer of tissue at the back of the inner eye that converts light images to nerve signals and sends them to the brain.Autologous Bone Marrow derived Mono Nuclear Stem Cell (BMMNCs) is used for this condition .

DETAILED DESCRIPTION:
This study will involve about 8 visits over 1½ years .Each participant will be enrolled in study as per inclusion and exclusion criteria .Informed consent will be taken from subject before including in study. Subject will be underwent for specific tests of the participant's vision and health. These visits may include visual exams, blood draw for laboratory testing, brief medical history and exam, and occasionally a questionnaire (survey), in addition to the visit for the surgical procedures. The primary outcome for this study will be a visual acuity score after one year of stem cell therapy .

Follow-up visits will be required regularly to determine the effectiveness of Autologous Bone Marrow derived Mono Nuclear Stem Cell (BMMNCs) in RP.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Diagnosis of retinitis pigmentosa
* willingness to undergo Bone marrow and umbilical cord derived Mesenchymal stem cell transplantation.
* To give an informed consent as well as sign the required Informed Consent Form (ICF) for the study.
* willingness to regularly visit the hospital / clinic for follow up during the follow up period / on prior agreed time points as per the protocol.

Exclusion Criteria:

* Positive test results for HIV and AIDS complex ,HCV (hepatitis C virus ), HbsAg and Syphilis
* Women who are pregnant or lactating
* Complications of diabetic retinopathy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
visual acuity | 1 YEAR
  Electronic Visual Acuity (EVA) technology

CONTACTS AND LOCATIONS:
Overall Officials: ANANT E BAGUL, MS ORTHO, Principal Investigator — Chaitanya Hospital
Locations (1):
- Chaitanya Hospital, Pune, Maharashtra, India